CLINICAL TRIAL: NCT00750880
Title: International Multi-Center Open Label Study to Evaluate the Safety, Tolerability and Efficacy of Tocilizumab in Patients With Active Rheumatoid Arthritis on Background Non-biologic DMARDs Who Have An Inadequate Response to Current Non-Biologic DMARD or Anti-TNF Therapy.
Brief Title: An Exploratory Study of Tocilizumab in Patients With Active Rheumatoid Arthritis (RA) and an Inadequate Response to Current Non-Biologic DMARDs and/or Anti-TNF Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA21573; 2008-000587-17
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv (60 minute infusion)

SUMMARY:
This open-label, single arm study will investigate the safety, tolerability and efficacy of tocilizumab monotherapy, or combination therapy with non-biologic disease modifying antirheumatic drugs (DMARDs), in patients with severe active RA. Patients will receive tocilizumab 8mg/kg iv as a 60 minute infusion every 4 weeks for a total of 6 infusions. The anticipated time on study treatment is 3-12 months, and the target sample size is >500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male and non-pregnant or nursing female patients >=18 years of age;
* body weight <=150kg;
* moderate to severe active RA (DAS28 >=3.2) of >=6 months duration;
* on >=1 non-biologic DMARDs at a stable dose for a period of >= 8 weeks prior to start of treatment;
* inadequate clinical response to a stable dose of non-biologic DMARD or anti-TNF therapy;
* if receiving oral corticosteroids, the dose must have been stable for at least 25 of 28 days prior to start of treatment.

Exclusion Criteria:

* major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following enrollment;
* rheumatic autoimmune disease other than RA;
* prior history of, or current inflammatory joint disease other than RA;
* functional class IV as defined by the ACR Classification of Functional Status in RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1681 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (249):
- Australia (8):
  - Canberra, Australian Capital Territory
  - Coffs Harbour, New South Wales
  - Kogarah, New South Wales
  - Parramatta Park, New South Wales
  - Adelaide, South Australia
  - Fitzroy, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
- Austria (7):
  - Graz
  - Graz-Eggenberg
  - Innsbruck
  - Linz
  - Salzburg
  - Stockerau
  - Vienna
- Belgium (11):
  - Aalst
  - Brussels
  - Edegem
  - Ghent
  - Hasselt
  - Heusy
  - Leuven
  - Liège
  - Merksem
  - Montignies S/ Sambre
  - Westmalle
- Canada (19):
  - Edmonton, Alberta
  - Lethbridge, Alberta
  - Kelowna, British Columbia
  - Nanaimo, British Columbia
  - Vancouver, British Columbia
  - Quispamsis, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Laval, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Rimouski, Quebec
  - Saint-Eustache, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan
- Czechia (6):
  - Bruntál
  - Ostrava
  - Prague
  - Sokolov
  - Uherské Hradiště
  - Zlín
- Denmark (5):
  - Aarhus
  - Copenhagen
  - Esbjerg
  - Hjørring
  - Silkeborg
- Finland (3):
  - Helsinki
  - Jyväskylä
  - Turku
- France (28):
  - Argenteuil
  - Aulnay-sous-Bois
  - Belfort
  - Bobigny
  - Bourg-en-Bresse
  - Caen
  - Cahors
  - Colmar
  - Corbeil-Essonnes
  - Dijon
  - La Rochelle
  - Liévin
  - Lomme
  - Lyon
  - Marseille
  - Montivilliers
  - Montpellier
  - Mulhouse
  - Paris
  - Pau
  - Poitiers
  - Reims
  - Roubaix
  - Saint-Brieuc
  - Strasbourg
  - Toulouse
  - Valence
  - Valenciennes
- Germany (11):
  - Berlin
  - Bielefeld
  - Freiburg im Breisgau
  - Greifswald
  - Hamburg
  - Jena
  - Kiel
  - Rostock
  - Saarbrücken
  - Wuppertal
  - Würzburg
- Greece (5):
  - Athens
  - Heraklion
  - Ioannina
  - Pátrai
  - Thessaloniki
- Hungary (5):
  - Budapest
  - Eger
  - Gyula
  - Szeged
  - Veszprém
- India (9):
  - Bangalore
  - Chennai
  - Hyderabad
  - Jaipur
  - Kolkata
  - Ludhiana
  - Mumbai
  - New Delhi
  - Pune
- Ireland (6):
  - Co Leitrim
  - Cork
  - Dublin
  - Galway
  - Limerick
  - Waterford
- Italy (12):
  - Arenzano
  - Legnano
  - Milan
  - Modena
  - Monserrato
  - Novara
  - Palermo
  - Pescara
  - Potenza
  - Roma
  - Siena
  - Varese
- Luxembourg, Luxembourg
- Netherlands (22):
  - 's-Hertogenbosch
  - Alkmaar
  - Amsterdam
  - Apeldoorn
  - Arnhem
  - Bergen op Zoom
  - Den Helder
  - Enschede
  - Flushing
  - Gorinchem
  - Gouda
  - Heerlen
  - Hilversum
  - Leeuwarden
  - Leidschendam
  - Nieuwegein
  - Nijmegen
  - Roosendaal
  - Rotterdam
  - Schiedam
  - Spijkenisse
  - The Hague
- Poland (3):
  - Krakow
  - Poznan
  - Wroclaw
- Portugal (4):
  - Almada
  - Coimbra
  - Lisbon
  - Porto
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Jeddah, Saudi Arabia
- Spain (30):
  - Alicante, Alicante
  - Elche, Alicante
  - Elda, Alicante
  - Almería, Almeria
  - Avilés, Avila
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Terrassa, Barcelona
  - Vic, Barcelona
  - Cáceres, Caceres
  - Cadiz, Cadiz
  - Jerez de la Frontera, Cadiz
  - Córdoba, Cordoba
  - Granada, Granada
  - Huesca, Huesca
  - A Coruña, La Coruña
  - Las Palmas de Gran Canaria, Las Palmas
  - León, Leon
  - Ponferrada, Leon
  - Lugo, Lugo
  - Madrid, Madrid
  - Málaga, Malaga
  - Murcia, Murcia
  - Ourense, Orense
  - Salamanca, Salamanca
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Santa Cruz de Tenerife, Tenerife
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Sweden (9):
  - Falun
  - Huddinge
  - Karlstad
  - Linköping
  - Malmo
  - Skövde
  - Stockholm
  - Uppsala
  - Västerås
- Switzerland (7):
  - Aarau
  - Basel
  - Fribourg
  - Geneva
  - Lucerne
  - Sankt Gallen
  - Zurich
- Turkey (Türkiye) (2):
  - Ankara
  - Istanbul
- United Kingdom (33):
  - Barnsley
  - Basingstoke
  - Bournemouth
  - Brighton
  - Burton-on-Trent
  - Bury Saint Edmonds
  - Cambridge
  - Cardiff
  - Chelmsford
  - Dudley
  - Dundee
  - Eastbourne
  - Gillingham
  - Harrogate
  - Huddersfield
  - Ipswich
  - Liverpool
  - Llantrisant
  - London
  - Londonderry
  - Maidstone
  - Metropolitan Borough of Wirral
  - Middlesbrough
  - Newcastle upon Tyne
  - Nottingham
  - Reading
  - Salford
  - Sheffield
  - Southport
  - Swindon
  - Torquay
  - Westcliffe-on-sea
  - Worthing

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab (TCZ) 8 Milligrams Per Kilogram (mg/kg): Participants received tocilizumab 8 mg/kg intravenously (IV) once every 4 weeks for 20 weeks (total of 6 infusions).
Period: Overall Study
Arm/Group | Tocilizumab (TCZ) 8 Milligrams Per Kilogram (mg/kg)
Started | 1681
Completed | 1466
Not Completed | 215
Not completed — Adverse Event | 76
Not completed — Death | 4
Not completed — Lack of Efficacy | 46
Not completed — Lost to Follow-up | 10
Not completed — Protocol Violation | 15
Not completed — Withdrawal by Subject | 33
Not completed — Physician Decision | 20
Not completed — Administrative | 11

BASELINE CHARACTERISTICS:
Population: Inten-to-Treat (ITT) population: all participants included in the study who received at least 1 dose of study medication.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg IV once every 4 weeks for 20 weeks (total of 6 infusions).
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1356
  Male | 325

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Achieved Low Disease Activity or Remission Based on Disease Activity Score Based on 28-Joints Count (DAS28) by Visit
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and Patient's Global Assessment of Disease Activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. Low disease activity was defined as DAS28 less than or equal to (≤)3.2 and remission was defined as DAS28 less than (<)2.6.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; no imputation of missing data was performed for this analysis.
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg iv infusions every 4 weeks for 24 weeks.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1677
percentage of participants
  Baseline, low disease activity (n=1677) | 1.1
  Baseline, DAS28 <2.6 (n=1677) | 0.2
  Week 4, low disease activity (n=1635) | 27.6
  Week 4, DAS28 <2.6 (n=1635) | 14.9
  Week 8, low disease activity (n=1594) | 49.2
  Week 8, DAS28 <2.6 (n=1594) | 32.6
  Week 12, low disease activity (n=1556) | 57.3
  Week 12, DAS28 <2.6 (n=1556) | 40.0
  Week 16, low disease activity (n=1509) | 64.7
  Week 16, DAS28 <2.6 (n=1509) | 48.4
  Week 20, low disease activity (n=1467) | 69.3
  Week 20, DAS28 <2.6 (n=1467) | 54.9
  Week 24, low disease activity (n=1455) | 69.9
  Week 24, DAS28 <2.6 (n=1455) | 56.8

2. Secondary Outcome: Time to Low Disease Activity or Remission Based on DAS28 - Number of Participants With an Event
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (mm/hr) and Patient's Global Assessment of Disease Activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. Low disease activity was defined as DAS28 ≤3.2 and remission was defined as DAS28 <2.6.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; Only population with complete DAS28 data were analyzed.
Measure: Number; unit: participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1665
participants
  Low disease activity | 1320
  DAS28 <2.6 | 1127

3. Secondary Outcome: Time to Low Disease Activity and Remission Based on DAS28 Score - Time to Event
Description: The time to low disease activity or remission was calculated as the number of days from study Day 1 to the first occurrence of low disease activity or remission. Participants who did not achieve low disease activity on or before Week 24 or who withdrew from the study prior to achieving low disease activity were considered censored. DAS28 calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (mm/hr) and Patient's Global Assessment of Disease Activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. Low disease activity defined as DAS28 ≤3.2 and remission defined as DAS28 <2.6.
Time Frame: Baseline,Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population with DAS28 ≤3.2
Measure: Median (Full Range); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1320
days
  Low disease activity (n=1320) | 63.0 [60.0 to 80.0]
  Remission (n=1127) | 112.0 [97.0 to 113.0]

4. Secondary Outcome: Percentage of Participants Achieving a Response by European League Against Rheumatism (EULAR) Response Category and Visit
Description: DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 ≤3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or change from baseline >0.6 to =<1.2 with DAS28 ≤5.1; non-responders: change from baseline ≤0.6 or change from baseline >0.6 and ≤1.2 with DAS28 >5.1. If the EULAR response could not be determined, it was set to 'No response'.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
percentage of participants
  Week 4, Good Response | 24.7
  Week 4, Moderate Response | 52.6
  Week 4, No Response | 22.7
  Week 8, Good Response | 44.7
  Week 8, Moderate Response | 40.8
  Week 8, No Response | 14.5
  Week 12, Good Response | 51.3
  Week 12, Moderate Response | 34.9
  Week 12, No Response | 13.7
  Week 16, Good Response | 57.0
  Week 16, Moderate Response | 27.5
  Week 16, No Response | 15.5
  Week 20, Good Response | 59.3
  Week 20, Moderate Response | 23.7
  Week 20, No Response | 17.0
  Week 24, Good Response | 59.6
  Week 24, Moderate Response | 23.8
  Week 24, No Response | 16.6

5. Secondary Outcome: DAS28 Scores by Visit
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (mm/hr) and Patient's Global Assessment of Disease Activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1677
units on a scale
  Baseline (n=1677) | 5.96 (1.201)
  Week 4 (n=1635) | 4.12 (1.451)
  Change at Week 4 (n=1631) | -1.84 (1.165)
  Week 8 (n=1594) | 3.35 (1.442)
  Change at Week 8 (n=1590) | -2.60 (1.336)
  Week 12 (n=1556) | 3.03 (1.431)
  Change at Week 12 (n=1552) | -2.92 (1.429)
  Week 16 (n=1509) | 2.80 (1.459)
  Change at Week 16 (n=1506) | -3.14 (1.464)
  Week 20 (n=1467) | 2.63 (1.428)
  Change at Week 20 (n=1463) | -3.14 (1.488)
  Week 24 (n=1455) | 2.52 (1.378)
  Change at Week 24 (n=1451) | -3.42 (1.438)

6. Secondary Outcome: Percentage of Participants Achieving an American College of Rheumatology 20 Percent (%), 50%, 70%, or 90% Improvement (ACR20/ACR50/ACR70/ACR90) by Visit
Description: ACR20, ACR50, ACR70, and ACR90 are defined as ≥20%, ≥50%, ≥70%, or ≥90% improvement, respectively, in: swollen joint count (SJC; 66 joints) and tender joint count (TJC; 68 joints) and ≥20%, ≥50%, ≥70%, or ≥90% improvement, respectively, in 3 of following 5 assessments: Patient's Global Assessment of Pain (visual analog scale [VAS]); Patient's Global Assessment of Disease Activity (VAS); Investigator/Physician's Global Assessment of Disease Activity (VAS); participant's assessment of disability measured by the Health Assessment Questionnaire Disability Index (HAQ-DI); or acute phase reactant (ESR or C-reactive protein [CRP]). Participants who did not have the required data to assess ACR status at a given visit were classified as non-responders.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
percentage of participants
  Week 4, ACR20 | 36.5
  Week 4, ACR50 | 10.5
  Week 4, ACR70 | 2.7
  Week 4, ACR90 | 0.3
  Week 8, ACR20 | 55.6
  Week 8, ACR50 | 26.9
  Week 8, ACR70 | 10.7
  Week 8, ACR90 | 2.2
  Week 12, ACR20 | 61.0
  Week 12, ACR50 | 36.3
  Week 12, ACR70 | 17.5
  Week 12, ACR90 | 4.8
  Week 16, ACR20 | 64.1
  Week 16, ACR50 | 40.2
  Week 16, ACR70 | 21.1
  Week 16, ACR90 | 5.8
  Week 20, ACR20 | 65.0
  Week 20, ACR50 | 44.4
  Week 20, ACR70 | 22.4
  Week 20, ACR90 | 6.7
  Week 24, ACR20 | 66.9
  Week 24, ACR50 | 46.6
  Week 24, ACR70 | 26.4
  Week 24, ACR90 | 8.7

7. Secondary Outcome: Time to Achieve ACR20, ACR50, ACR70 and ACR90 Response - Number of Participants With an Event
Description: ACR20, ACR50, ACR70, and ACR90 are defined as ≥20%, ≥50%, ≥70%, or ≥90% improvement, respectively, in: swollen joint count (SJC; 66 joints) and tender joint count (TJC; 68 joints) and ≥20%, ≥50%, ≥70%, or ≥90% improvement, respectively, in 3 of following 5 assessments: Patient's Global Assessment of Pain (VAS); Patient's Global Assessment of Disease Activity (VAS); Investigator/Physician's Global Assessment of Disease Activity (VAS); participant's assessment of disability measured by the HAQ-DI; or acute phase reactant (ESR or CRP).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
participants
  ACR20 | 1431
  ACR50 | 1075
  ACR70 | 659
  ACR90 | 232

8. Secondary Outcome: Time to Achieve ACR20, ACR50, ACR70 and ACR90 Response
Description: ACR20, ACR50, ACR70, and ACR90 are defined as ≥20%, ≥50%, ≥70%, or ≥90% improvement, respectively, in: swollen joint count (SJC; 66 joints) and tender joint count (TJC; 68 joints) and ≥20%, ≥50%, ≥70%, or ≥90% improvement, respectively, in 3 of following 5 assessments: Patient's Global Assessment of Pain (VAS); Patient's Global Assessment of Disease Activity (VAS); Investigator/Physician's Global Assessment of Disease Activity (VAS); participant's assessment of disability measured by the HAQ-DI; or acute phase reactant (ESR or CRP). Time to ACR response was calculated as the number of days from day 1 of study to the date of first achievement of ACR response. Data represent median time for responders only.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; only participants with a response (ACR20/ACR50/ACR70/ACR90) were included in the analysis. n=number of participants with a response for the specified parameter
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1431
days
  ACR20 (n=1431) | 57.0 [22 to 197]
  ACR50 (n=1075) | 84.0 [23 to 243]
  ACR70 (n=659) | 90.0 [25 to 238]
  ACR90 (n=232) | 113.0 [27 to 197]

9. Secondary Outcome: Swollen Joint Count by Visit
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 66. A negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; missing data were handled using the LOCF approach.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
swollen joints
  Baseline | 12.76 (9.183)
  Week 4 | 9.24 (10.371)
  Change at Week 4 | -3.52 (10.882)
  Week 8 | 6.56 (8.799)
  Change at Week 8 | -6.20 (10.597)
  Week 12 | 5.62 (8.324)
  Change at Week 12 | -7.14 (10.737)
  Week 16 | 5.24 (8.441)
  Change at Week 16 | -7.52 (11.114)
  Week 20 | 4.77 (8.150)
  Change at Week 20 | -7.99 (11.130)
  Week 24 | 4.60 (8.216)
  Change at Week 24 | -8.16 (11.179)

10. Secondary Outcome: Tender Joint Count by Visit
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 68. A negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; missing data were handled using the last observation carried forward (LOCF) approach.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
tender joints
  Baseline | 22.82 (15.019)
  Week 4 | 16.55 (15.024)
  Change at Week 4 | -6.27 (13.384)
  Week 8 | 12.21 (13.227)
  Change at Week 8 | -10.61 (13.960)
  Week 12 | 10.47 (12.831)
  Change at Week 12 | -12.35 (14.611)
  Week 16 | 9.75 (12.372)
  Change at Week 16 | -13.06 (14.876)
  Week 20 | 9.31 (12.326)
  Change at Week 20 | -13.51 (15.312)
  Week 24 | 8.74 (12.115)
  Change at Week 24 | -14.08 (15.520)

11. Secondary Outcome: Patient's Global Assessment of Disease Activity by Visit
Description: The participant's global assessment of disease activity is assessed on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line=0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme=100 mm, as "maximum disease activity" (maximum arthritis disease activity). The line was marked by the participant and the distance from the left edge was recorded. A negative change from baseline indicated improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1677
mm
  Baseline (n=1677) | 62.52 (21.192)
  Week 4 (n=1653) | 47.20 (23.945)
  Change at Week 4 (n=1649) | -15.32 (23.852)
  Week 8 (n=1610) | 37.95 (24.377)
  Change at Week 8 (n=1606) | -24.52 (25.972)
  Week 12 (n=1569) | 33.27 (23.474)
  Change at Week 12 (n=1565) | -28.98 (25.885)
  Week 16 (n=1525) | 30.92 (23.720)
  Change at Week 16 (n=1522) | -31.42 (26.213)
  Week 20 (n=1488) | 28.74 (22.948)
  Change at Week 20 (n=1484) | -33.42 (26.160)
  Week 24 (n=1472) | 26.68 (22.070)
  Change at Week 24 (n=1468) | -35.53 (25.558)

12. Secondary Outcome: Physician's Global Assessment of Disease Activity by Visit
Description: The physician's global assessment of disease activity is assessed on a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line=0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme=100 mm as "maximum disease activity" (maximum arthritis disease activity). The physician marked the line and the distance from the left edge was recorded. A negative change from baseline indicated improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1675
mm
  Baseline (n=1675) | 58.82 (17.886)
  Week 4 (n=1645) | 39.79 (19.858)
  Change at Week 4 (n=1640) | -18.93 (20.126)
  Week 8 (n=1605) | 30.01 (18.671)
  Change at Week 8 (n=1601) | -28.65 (21.190)
  Week 12 (n=1567) | 25.71 (18.217)
  Change at Week 12 (n=1563) | -32.72 (21.295)
  Week 16 (n=1525) | 23.17 (17.646)
  Change at Week 16 (n=1521) | -35.49 (21.636)
  Week 20 (n=1482) | 21.18 (17.064)
  Change at Week 20 (n=1478) | -37.33 (21.855)
  Week 24 (n=1459) | 19.53 (17.183)
  Change at Week 24 (n=1455) | -39.10 (21.984)

13. Secondary Outcome: Patient's Global Assessment of Pain by Visit
Description: The participants assessed their pain using a 0 to 100 mm horizontal VAS. The left-hand extreme of the line=0 mm, and is described as "no pain" and the right-hand extreme=100 mm as "unbearable pain". The participant marked the line and the distance from the left edge was recorded. A negative change from baseline indicated improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1675
mm
  Baseline (n=1675) | 57.51 (22.582)
  Week 4 (n=1654) | 43.10 (23.563)
  Change at Week 4 (n=1648) | -14.41 (23.441)
  Week 8 (n=1612) | 34.93 (23.711)
  Change at Week 8 (n=1606) | -22.51 (25.138)
  Week 12 (n=1572) | 31.02 (23.342)
  Change at Week 12 (n=1566) | -26.21 (26.036)
  Week 16 (n=1525) | 28.56 (23.016)
  Change at Week 16 (n=1521) | -28.59 (26.079)
  Week 20 (n=1489) | 26.76 (22.456)
  Change at Week 20 (n=1483) | -30.29 (26.417)
  Week 24 (n=1473) | 24.90 (21.398)
  Change at Week 24 (n=1468) | -32.13 (25.925)

14. Secondary Outcome: C-Reactive Protein by Visit
Description: The test for CRP (mg per deciliter [mg/dL]) is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
mg/dL
  Baseline (n=1681) | 1.94 (2.775)
  Week 4 (n=1649) | 0.52 (1.834)
  Change at Week 4 (n=1649) | -1.40 (2.243)
  Week 8 (n=1613) | 0.36 (1.372)
  Change at Week 8 (n=1613) | -1.59 (2.474)
  Week 12 (n=1571) | 0.28 (1.247)
  Change at Week 12 (n=1571) | -1.63 (2.532)
  Week 16 (n=1525) | 0.23 (0.798)
  Change at Week 16 (n=1525) | -1.70 (2.655)
  Week 20 (n=1481) | 0.23 (1.078)
  Change at Week 20 (n=1481) | -1.68 (2.573)
  Week 24 (n=1448) | 0.19 (0.802)
  Change at Week 24 (n=1448) | -1.74 (2.608)

15. Secondary Outcome: Erythrocyte Sedimentation Rate by Visit
Description: ESR (mm/hr) is a blood test used to monitor therapy in inflammatory diseases such as rheumatoid arthritis (RA) and reflects acute phase reactant levels. Active disease in RA is defined by an ESR greater than 30 mm/hr. Change from baseline is computed as the value at each week minus the baseline value. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
mm/hr
  Baseline (n=1681) | 39.20 (26.843)
  Week 4 (n=1642) | 13.13 (16.468)
  Change at Week 4 (n=1642) | -26.07 (21.863)
  Week 8 (n=1603) | 10.26 (14.935)
  Change at Week 8 (n=1603) | -28.93 (23.945)
  Week 12 (n=1567) | 8.97 (12.527)
  Change at Week 12 (n=1567) | -30.02 (24.543)
  Week 16 (n=1520) | 8.39 (12.230)
  Change at Week 16 (n=1520) | -30.43 (24.703)
  Week 20 (n=1474) | 7.81 (11.653)
  Change at Week 20 (n=1474) | -31.01 (24.648)
  Week 24 (n=1463) | 7.90 (11.485)
  Change at Week 24 (n=1463) | -31.01 (24.796)

16. Secondary Outcome: HAQ-DI Scores by Visit
Description: HAQ-DI includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0 (equals)=without difficulties; 1=with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1673
units on a scale
  Baseline (n=1673) | 1.49 (0.637)
  Week 4 (n=1648) | 1.27 (0.665)
  Change at Week 4 (n=1641) | -022 (0.448)
  Week 8 (n=1607) | 1.12 (0.677)
  Change at Week 8 (n=1600) | -0.37 (0.511)
  Week 12 (n=1570) | 1.03 (0.684)
  Change at Week 12 (n=1562) | -0.46 (0.553)
  Week 16 (n=1524) | 0.99 (0.690)
  Change at Week 16 (n=1517) | -0.50 (0.566)
  Week 20 (n=1483) | 0.95 (0.687)
  Change at Week 20 (n=1476) | -0.53 (0.573)
  Week 24 (n=1459) | 0.92 (0.697)
  Change at Week 24 (n=1451) | -0.57 (0.585)

17. Secondary Outcome: Short Form-36 (SF-36) Physical Functioning Domain Scores by Visit
Description: The SF-36 covers 8 health dimensions including 4 physical subscales (physical function, role-physical, bodily pain, and general health) and 4 mental subscales (vitality, social function, role-emotional, and mental health). The scores range from a minimum of 0 to a maximum of 100, with a higher score indicating better quality of life. Improvements of >3 points were considered clinically meaningful.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1671
units on a scale
  Baseline (n=1671) | 31.39 (9.813)
  Week 4 (n=1647) | 34.17 (10.398)
  Change at Week 4 (1639) | 2.79 (8.064)
  Week 8 (n=1608) | 36.39 (10.829)
  Change at Week 8 (n=1598) | 4.95 (9.088)
  Week 12 (n=1573) | 37.69 (11.096)
  Change at Week 12 (n=1564) | 6.19 (9.751)
  Week 16 (n=1529) | 38.41 (11.139)
  Change at Week 16 (n=1521) | 6.89 (9.850)
  Week 20 (n=1487) | 39.21 (11.123)
  Change at Week 20 (n=1479) | 7.66 (10.306)
  Week 24 (n=1465) | 39.52 (11.302)
  Change at Week 24 (n=1457) | 7.92 (10.211)

18. Primary Outcome: Percentage of Participants With Adverse Events (AEs): Overall Summary
Description: Percentage of participants with AEs, serious AEs (SAEs), related AEs, related SAEs, severe AEs, with AEs leading to withdrawal or dose modification, with infection, serious infection, infusion reactions, infusion reactions during an infusion, infusion reactions within 24 hours of an infusion, major adverse cardiac event (MACE), or death.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: Safety population: all participants included in the study who received at least 1 dose of study medication and who had at least 1 postbaseline assessment of safety (post-baseline laboratory data, vital signs, or adverse events). number (n) equals (=) number of participants analyzed for the parameter within the specific population.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1681
percentage of participants
  Any AE | 77.4
  Related AE | 58.4
  Severe AE | 7.8
  SAE | 7.8
  Related SAE | 3.5
  AE leading to withdrawal | 5.1
  AE leading to dose modification | 10.8
  Infection | 35.3
  Serious infection | 2.1
  Any infusion reaction (during or within 24 hours) | 17.3
  Infusion reaction during infusion | 6.7
  Infusion reaction within 24 hours of infusion | 12.6
  MACE | 0.4
  Death | 0.2

19. Secondary Outcome: Percentage of Participants With HAQ-DI Clinical Remission and Clinically Meaningful Improvement By Visit
Description: The HAQ-DI scale ranges from 0 to 3, where higher scores represent higher disease activity. A score of <0.5 represents clinical remission. A participant achieves a clinically meaningful improvement in HAQ-DI if they had a reduction from baseline of ≥0.22.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1673
percentage of participants
  Baseline, Remission (n=1673) | 5.9
  Week 4, Remission (n=1648) | 12.6
  Week 4, Clinically meaningful improvement (n=1641) | 47.7
  Week 8, Remission (n=1607) | 19.0
  Week 8, Clinically meaningful improvement (n=1600) | 60.4
  Week 12, Remission (n=1570) | 23.9
  Week 12 Clinically meaningful improvement (n=1562) | 65.7
  Week 16, Remission (n=1524) | 26.4
  Week 16 Clinically meaningful improvement (n=1517) | 68.7
  Week 20, Remission (n=1483) | 28.1
  Week 20 Clinically meaningful improvement (n=1476) | 70.6
  Week 24, Remission (n=1459) | 31.5
  Week 24, Clinically meaningful improvement(n=1451) | 72.7

20. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score by Visit
Description: FACIT-Fatigue is a 13-item questionnaire; participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the participant's health status.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 1674
units on a scale
  Baseline (n=1674) | 25.91 (11.262)
  Week 4 (n=1647) | 30.95 (11.133)
  Change at Week 4 (n=1640) | 5.01 (8.916)
  Week 8 (n=1611) | 33.51 (10.865)
  Change at Week 8 (n=1605) | 7.50 (10.036)
  Week 12 (n=1573) | 34.98 (11.069)
  Change at Week 12 (n=1568) | 8.86 (10.463)
  Week 16 (n=1529) | 35.78 (10.959)
  Change at Week 16 (n=1524) | 9.68 (10.890)
  Week 20 (n=1488) | 36.45 (10.848)
  Change at Week 20 (n=1483) | 10.31 (10.947)
  Week 24 (n=1466) | 36.92 (10.823)
  Change at Week 24 (n=1461) | 10.76 (10.934)

ADVERSE EVENTS:
Time Frame: AE evaluation was done from the day of screening till the end of study at Week 24.
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 131/1681
Other Adverse Events (participants affected / at risk) | 370/1681
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=1681)
Pneumonia (Infections and infestations) | 6
Erysipelas (Infections and infestations) | 5
Bursitis infective (Infections and infestations) | 2
Alveolar osteitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bordetella infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Joint tuberculosis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Meningitis viral (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Postoperative abscess (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Scrotal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Tendon injury (Injury, poisoning and procedural complications) | 2
Tendon rupture (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Sciatica (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Chest pain (General disorders) | 4
Ill-defined disorder (General disorders) | 1
Infusion related reaction (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deep vein thrombosis (Vascular disorders) | 2
Aortic dissection (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Rheumatoid vasculitis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Arteriospasm coronary (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Depression (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Corneal perforation (Eye disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Blood pressure increased (Investigations) | 1
Testicular cyst (Reproductive system and breast disorders) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=1681)
Nasopharyngitis (Infections and infestations) | 116
Blood cholesterol increased (Investigations) | 105
Hypercholesterolaemia (Metabolism and nutrition disorders) | 101
Headache (Nervous system disorders) | 92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.